CLINICAL TRIAL: NCT00502827
Title: An Innovative Telephone Intervention for HIV-Positive Smokers
Brief Title: Smoking Cessation for HIV/AIDS Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2003-0784; NCI-2012-02109 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-07-16; First posted 2007-07-18 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Human Immunodeficiency Virus
Keywords: Human Immunodeficiency Virus; HIV positive; HIV Positive Smokers; AIDS; Cell Phone Intervention; CPI; Smoking Cessation; Interview
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Seropositivity; Smoking Cessation | interventions — cyclopropapyrroloindole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Recommended Standard of Care (Other): Recommended Standard of Care (RSOC) = Physician Advice + Written Materials
  Interventions: Other: Recommended Standard of Care
- RSOC + Cell Phone Intervention (Other): Recommended Standard of Care (RSOC) + Cell Phone Intervention
  Interventions: Behavioral: Cell Phone Intervention; Other: Recommended Standard of Care

INTERVENTIONS:
Behavioral: Cell Phone Intervention — Study participants called on a cell phone 11 times over course of a 12 - 13 week period, during 10 minute calls questions asked about smoking and quitting smoking.
  Other Names: CPI
  Arms: RSOC + Cell Phone Intervention
Other: Recommended Standard of Care — Advice from your physician to stop smoking and written materials designed to help you quit smoking.
  Other Names: RSOC

SUMMARY:
The goal of this research study is to look at treatments that may help individuals who have HIV/AIDS to stop smoking.

DETAILED DESCRIPTION:
If you agree to take part in this study, researchers will first do a test to learn what the CO level of your blood is. To do this test, you will be asked to blow into a cardboard tube. If the test finds that you are ineligible, you will not be able to continue on this study.

If you are found to be eligible, you will be enrolled in this study and asked to complete an interview that should last about 1 hour. During this interview, you will be asked basic questions, such as your age, education level, and smoking history. You will also be asked questions about your mood, quality of life, and stress. You will then be asked to complete a short test that involves completing some basic tasks, such as remembering several words and drawing a simple shape. This test, which will take about 2-5 minutes to complete, is used to measure attention and concentration.

You will then be randomly assigned (as in the toss of a coin) to one of two treatment groups. There is an equal chance of being assigned to either group.

If you are assigned to Group 1, you will receive advice from your physician/provider to stop smoking and written materials designed to help you quit smoking.

If you are assigned to Group 2, you will receive the advice from your physician/provider to quit smoking and the written materials, but you also be given a cell phone and be called 11 times over the course of an 12 to 13 week period. During these calls, which will last about 10 minutes, you will be asked to talk about smoking and quitting smoking. Access to a hotline number that you can call to speak with a counselor about quitting smoking will also be given to you if you are assigned to group 2. Participants in Group 1 will not get the number to the hotline. There is a limited number of prepaid minutes on the phone, so participants who receive a cell phone should make an effort to save enough minutes to complete this study.

You will be asked to complete three more interviews about 3-, 6-, and 12-months after the first interview. During these interviews, you will again be asked questions about your smoking behavior, mood, quality of life, and stress. All three of these interviews will take about one hour to complete. Your participation in this study will be complete after the 12-month interview.

Lost, stolen, or broken cell phones will not be replaced, but participants will remain on study.

This is an investigational study. Up to 705 participants will take part in this research study. All participants will be enrolled at Thomas Street Clinic.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-positive
2. 18 years of age or older
3. Current, regular smoker (> 5 cigarettes per day for the past 30 days, breath CO of > 7ppm)
4. English or Spanish speaking
5. Able to provide written informed consent to participate
6. Willing to set a quit date within 1 week of baseline assessment

Exclusion Criteria:

1. Physician deemed ineligibility based on medical (HIV related or other condition) or psychiatric condition
2. Current participation in another smoking cessation program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 706 (Actual)
Dates: Start 2004-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Proportion of participants in the two intervention groups who are abstinent as measured by point prevalence | 1 year after quit date

CONTACTS AND LOCATIONS:
Overall Officials: Damon Vidrine, MS, DRPH, BA, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Thomas Street Clinic, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Mdege ND, Shah S, Dogar O, Pool ER, Weatherburn P, Siddiqi K, Zyambo C, Livingstone-Banks J. Interventions for tobacco use cessation in people living with HIV. Cochrane Database Syst Rev. 2024 Aug 5;8(8):CD011120. doi: 10.1002/14651858.CD011120.pub3. PMID 39101506
- [Derived] Buchberg MK, Gritz ER, Kypriotakis G, Arduino RC, Vidrine DJ. The role of BMI change on smoking abstinence in a sample of HIV-infected smokers. AIDS Care. 2016;28(5):603-7. doi: 10.1080/09540121.2015.1120854. Epub 2015 Dec 15. PMID 26666313
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org